CLINICAL TRIAL: NCT00066638
Title: A Phase 2 Study of Depsipeptide in Relapsed/Refractory Multiple Myeloma
Brief Title: FR901228 in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03005; NCI-2012-03005 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-5996; 0403-765 (Other: Montefiore Medical Center - Moses Campus); 5996 (Other: CTEP); N01CM62204 (NIH); P30CA013330 (NIH)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2012-12

CONDITIONS: DS Stage II Plasma Cell Myeloma; DS Stage III Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — romidepsin

ARMS (1):
- Treatment (romidepsin) (Experimental): Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who achieve a stable plateau (stable paraprotein levels or urine protein excretion over 3 consecutive determinations at least 4 weeks apart) may receive maintenance therapy comprising FR901228 IV on days 1 and 15, with courses repeating every 28 days.
  Interventions: Drug: Romidepsin; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Romidepsin — Given IV
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy such as FR901228 use different ways to stop cancer cells from dividing so they stop growing or die. Phase II trial to study the effectiveness of FR901228 in treating patients who have relapsed or refractory multiple myeloma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and efficacy of depsipeptide in patients with refractory or relapsed multiple myeloma (MM).

OUTLINE: This is a multicenter study.

Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who achieve a stable plateau (stable paraprotein levels or urine protein excretion over 3 consecutive determinations at least 4 weeks apart) may receive maintenance therapy comprising FR901228 IV on days 1 and 15, with courses repeating every 28 days.

PROJECTED ACCRUAL: A total of 21-50 patients will be accrued for this study within 5-12.5 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed stage IIa or IIIa multiple myeloma
* Patient has progressive disease and has had 1, 2, 3, or 4 prior lines of therapy
* Bilirubin < 2.0 mg/dL
* SGOT/SGPT =< 2.5 X institutional upper limit of normal
* Serum creatinine =< 1.5 mg/dl OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Karnofsky Performance Status equal or greater than 70%; KPS 60% will be allowed if reduced KPS is due to advanced skeletal disease
* Measurable disease as defined by serum M protein >= 1.0 gm/dl measured by serum protein electrophoresis or free light chain measurement, or quantitative immunoglobulins and/or urinary M protein excretion >= 200 mg/24 hrs
* Ejection fraction >= 50% and normal baseline EKG tracing
* No known central nervous system abnormality including neoplastic, vascular, inflammatory, degenerative or epilepsy
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Patients in whom cytopenias are considered to be due to myeloma marrow infiltration will be allowed as long as they meet the following criteria:

  * Bone marrow biopsy displaying >= normal cellularity for age and >= 50% involvement by myeloma
  * ANC > 1,000 and platelets > 50,000
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign written informed consent

Exclusion Criteria:

* Administration of chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to enrollment or unresolved adverse events due to agents administered more than 4 weeks earlier
* Prior treatment with a histone deacetylase inhibitor
* Patients may not be receiving any other investigational agent
* History of second cancer (except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free >= 5 years)
* Non secretory disease or plasma cell leukemia (> 2000 circulating plasma cells/uL)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to depsipeptide
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with left ventricular hypertrophy or history of arrhythmias including atrial fibrillation, myocardial infarction or congestive heart failure; patients may not be taking hydrochlorothiazides
* Patients that are pregnant or lactating will be excluded from this trial
* Known HIV positivity; patients infected with the HIV virus will be excluded from this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-06; Primary Completion 2007-05 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Response rate (complete response [CR] or partial response [PR]) | Up to 8 years
Event free survival | Up to 8 years

SECONDARY OUTCOMES:
Gene array parameters | Up to 8 years
  This analysis will be descriptive and will compare patterns of gene and phenotype expression pre and post therapy.
Immunochemistry parameters | Up to 8 years
  This analysis will be descriptive and will compare patterns of gene and phenotype expression pre and post therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Niesvizky-Iszaevich, Principal Investigator — Montefiore Medical Center - Moses Campus
Locations (1):
- Montefiore Medical Center - Moses Campus, The Bronx, New York, United States